CLINICAL TRIAL: NCT01104441
Title: Cardiovascular Events at One Year of Patients Hospitalized for Critical Limb Ischaemia and Aspirin Resistant Using the VerifyNow®. Aspirin Resistance and Prognosis of Patients With Critical Limb Ischaemia
Brief Title: Aspirin Resistance and Prognosis of Patients With Critical Limb Ischaemia
Acronym: Aspirine
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I08022
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2011-05

CONDITIONS: Aspirin Resistance
Keywords: critical limb ischaemia; Aspirin resistance
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acetylsalicylic acid (Aspirin, ASA) is the most widely prescribed drug used in primary and secondary prevention of cardiovascular disease. However, aspirin resistance has been described, mostly in cardiac patients and is an independent predictive factor for a poor survival. Two frequent conditions in patients with cardiovascular diseases, diabetes and hypercholesterolemia, are also considered as risk factors for aspirin resistance. Among patients with peripheral arterial disease, those with critical limb ischemia have the worst cardiovascular prognosis. At one year, 23% are dead, 25% have a major cardiovascular event and 25% have a major amputation (which can be combined). Aspirin resistance is poorly studied in these patients, and to our knowledge no study has been made to assess the prognosis value of aspirin resistance on cardiovascular outcomes in critical limb ischaemia patients.

Hospitalized critical limb ischaemia patients will be tested for aspirin resistance using the bed-side point of care VerifyNow®, and will be followed during one year, including death, fatal and non-fatal acute coronary syndromes, cardiac decompensation, stroke, and major amputation.

ELIGIBILITY:
Inclusion Criteria:

* any adult patient hospitalized for critical limb ischaemia and already treated by aspirin for at least 4 days before the VerifyNow® test. Critical limb ischemia is defined by the TASC II criteria : chronic ischemic rest pain, ulcers or gangrene attributable to objectively proven arterial occlusive disease, confirmed by an ankle pressure subordinate or equal 50 mmHg and a toe pressure subordinate or equal 30 mmHg, or a transcutaneous oxygen tension subordinate or equal 30 mmHg

Exclusion Criteria:

* non observance to aspirin treatment, other drugs that could interact with platelets (NSAIDs, other anti-platelet agents), other peripheral vascular disease status than critical limb ischemia, acute limb ischemia, platelet number lower than 100 000/mm3, hematocrit lower than 29%, known primary hemostasis disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized for critical limb ischaemia and aspirin resistant using the VerifyNow®.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac events (MACE) including death, acute coronary syndromes, cardiac decompensation, stroke, major amputations. | 2 years

SECONDARY OUTCOMES:
major amputations, death | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - UH Bordeaux, Bordeaux
  - UH Toulouse, Toulouse